CLINICAL TRIAL: NCT04291820
Title: Anaesthesiology Management and the Impact on Emergenece Delirium Incidence in Paediatric Patients Undergoing Adenoidectomy or Adenoidectomy With Frenulum Dicsision a/or Microotoscopy: Randomized Controlled Trial
Brief Title: Impact of Anaesthesiology Management on Paediatric Emergence Delirium Incidence
Acronym: AnaPed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KDAR SUP 2020
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Emergence Delirium
Keywords: Delirium; Emergence delirium; Paediatric patient; Anaesthesia
MeSH Terms: conditions — Emergence Delirium; Delirium | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: A prospective interventional single-blind randomized trial
Who Masked: Outcomes Assessor
Masking Description: The participants will be blinded by the arm inclusion. The outcomes will be measured by the blinded nurse in the PACU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous induction with desflurane maintenance (Experimental): The EMLA patch will be removed, and intravenous induction with propofol + opioid will be performed. The anaesthesia will be maintained with desflurane according to the levels of Bispectral index (BIS). Neuromuscular blockade is optional based on operator decision.
  Interventions: Procedure: Intravenous induction and desflurane anaesthesia maintenance
- Inhalation induction with sevoflurane,sevoflurane maintenance (Active Comparator): The EMLA patch will be removed, and inhalation induction with the sevoflurane will be performed. After peripheral vein cannulation, the opioid will be administered. The neuromuscular blockade is optional based on operator decision. Anaesthesia will be maintained with sevoflurane according to the set BIS levels.
  Interventions: Procedure: Inhalation induction with sevoflurane and anaesthesia maintenance with sevoflurane

INTERVENTIONS:
Procedure: Intravenous induction and desflurane anaesthesia maintenance — Anaesthesia will be inducted with intravenous propofol + opioid and maintained with desflurane according to the BIS levels
  Arms: Intravenous induction with desflurane maintenance
Procedure: Inhalation induction with sevoflurane and anaesthesia maintenance with sevoflurane — Anaesthesia will be inducted with sevoflurane and maintained with sevoflurane according to the BIS levels
  Arms: Inhalation induction with sevoflurane,sevoflurane maintenance

SUMMARY:
Postoperative emergence delirium (ED) is a severe postoperative complication in paediatric anaesthesia. ED is defined as a state with psychomotor disturbance, perception disorder and state of excitation and anxiety. The incidence of ED in paediatric patients can be up to 80%. ED is associated with the increased morbidity of paediatric patients in the postoperative period. One of the potential triggers of ED is sevoflurane. Currently, there are only limited data about comparing the influence of anesthesiologic management on the ED incidence. The possible ED reduction could lead to reduced stay in a post-anaesthesia care unit (PACU), postoperative nausea and vomiting (PONV) incidence and the overall reduction of the postoperative adverse events incidence together with the higher satisfaction and the patients and the legal guardians.

DETAILED DESCRIPTION:
This prospective randomized interventional single-blind study aims to compare the influence of the anaesthesiology management no the incidence of ED in the postoperative period in paediatric patients. Elective paediatric patients (2-10 years) scheduled for the planned adenoidectomy or adenoidectomy + micro-otoscopy/adenoidectomy + frenulum linguae discission will be included in the trial after signed informed consent form the legal guardian. In all patients, the 2 Eutectic Mixture of Local Anesthetics (EMLA) patch will be applied on the predefined skin area ( visible vein for venepuncture) between 45 minutes to 60 minutes before anaesthesia. The patients will be randomized at the operating theatre (allocation 1:1) into the experimental group (intravenous induction with propofol + opioid and anaesthesia maintenance according to this set bispectral index value with desflurane) and the control group (inhalation induction with sevoflurane mixed with air and oxygen and anaesthesia maintenance with sevoflurane). The primary aim of the study will be the incidence of ED defined by The Pediatric Anesthesia Emergence Delirium (PAED) scale, which will be measured at the , at the admission to PACU and in the 5th, 10th, 15th, 30th minute and at the moment of dismission from PACU. The secondary aim will be the time to oral intake (from the end of the surgery), the incidence of adverse events (PONV, bradycardia, hypotension), the need for concomitant medication (analgesic medication, sedative medication, antiemetic medication).

ELIGIBILITY:
Inclusion Criteria:

* age between 2-10 years
* signed informed consent
* paediatric patient for elective adenoidectomy, or adenoidectomy with micro-otoscopy and/or frenulum discission

Exclusion Criteria:

* allergy and hypersensitivity on local anaesthetics in EMLA patch, general anaesthetics, or soya beans or peanuts
* venepuncture refusal · neuromuscular disorder with the contraindication of inhalation anaesthetics

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergence delirium incidence | postoperative period, up to 1 hour postoperatively
  The incidence of emergence delirium based on PAED score

SECONDARY OUTCOMES:
Time to first oral intake | postoperative period, up to 1 hour postoperatively
  The interval between the end of surgery and first oral intake will be measured
Adverse events incidence | postoperative period, up to 1 hour postoperatively
  The adverse events in the postoperative period will be evaluated - postoperative nausea and vomiting, bradycardia, hypotension, anxiety
The need for concomitant medication in PACU | postoperative period, up to 1 hour postoperatively
  The need for concomitant medication in PACU - analgesic, sedative, antiemetic medication

CONTACTS AND LOCATIONS:
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided